CLINICAL TRIAL: NCT05731323
Title: A Pharmacokinetic Study of Adjunctive D-cycloserine to Intermittent Theta Burst Stimulation in Major Depressive Disorder
Brief Title: D-Cycloserine+iTBS PK Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB22-0547
Record Dates: First submitted 2022-11-02; First posted 2023-02-16 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Cycloserine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- D-Cycloserine (Experimental): Prior to initiating TMS therapy, participants will orally ingest a capsule containing 100mg of the antibiotic d-cycloserine.
  During TMS therapy, participants will orally ingest a capsule containing a weight-based dose of the antibiotic d-cycloserine (dosed 25mg/17.5kg body weight) daily (Monday-Friday) for 4 weeks of rTMS treatment (20 sessions).
  Interventions: Drug: D-cycloserine; Device: Transcranial Magnetic Stimulator

INTERVENTIONS:
Drug: D-cycloserine — Daily oral D-cycloserine dosed 25mg/17.5kg body weight during TMS treatment days (20 days).
  Other Names: Seromycin
Device: Transcranial Magnetic Stimulator — Repetitive Transcranial magnetic stimulation (rTMS) will be delivered using a MagPro X100 device with B70 coil and the intermittent theta burst (iTBS) protocol to the left dorsolateral prefrontal cortex. Participants will receive daily treatments (Monday-Friday) over four weeks.

SUMMARY:
Background & Rationale: Major Depressive Disorder (MDD) is a common and debilitating illness that that commonly does not respond to conventional treatments. Transcranial magnetic stimulation (TMS) and intermittent theta-burst stimulation (iTBS) are non-invasive neurostimulation treatments for depression that are Health Canada approved. These work by generating magnetic fields outside of the body to change the activity of brain cells to change how the brain works. They have a very favorable profile, with many patients experiencing improvement with minimal side effects.

The investigators recently completed a study pairing iTBS with an FDA approved medication that was chosen because it might enhance iTBS improvements. This medication is called D-cycloserine, an old antibiotic that is rarely used in modern times. Years after it stopped being useful as an antibiotic, scientists recognized other properties that the molecule has, and it is some of these that make it interesting to pair with iTBS. When the investigators did so, they found that compared to iTBS with a placebo, participants who received iTBS+D-cycloserine were more likely to benefit from treatment.

In this original study, all participants received a fixed dose of 100mg daily. This means that people of very different sizes could have had different drug levels, and the investigators do not know how that impacted outcomes. With this study, there will be no placebo condition because the purpose is to understand whether dosing according to weight matters.

Research Question and Objectives: To describe the pharmacokinetic profile of 100mg oral D-cycloserine and weight-based oral D-cycloserine dosed 25mg/17.5kg among individuals with depression undergoing non-invasive intermittent theta-burst stimulation to the left dorsolateral prefrontal cortex (DLPFC) in Major Depressive Disorder.

DETAILED DESCRIPTION:
Methods: An open-label study of D-cycloserine (DCS) pharmacokinetics will be performed in patients undergoing iTBS to the left DLPFC as a treatment for Major Depressive Disorder. Twelve patients (males and females aged 18-65, with a score ≥18 on the Hamilton Rating Scale for Depression-17 items, and stable pharmacological and psychological regimens) with an acute Major Depressive Episode will be recruited. Bloodwork and an echocardiogram will be obtained prior to the initiation of the study, and enrollment in the study will be contingent on normal lab results.

Prior to initiating iTBS treatment, participants will receive one oral dose of 100mg DCS. A pharmacokinetic curve will be generated from D-Cycloserine levels obtained at 6 timepoints; pre-ingestion, +30 mins, + 60 mins, + 90mins, +120mins and +24 hrs.

Participants will receive iTBS daily for 4 weeks (20 sessions). All participants will be provided with weight-based dosing of DCS to take 120 minutes prior to each iTBS session. Serum levels of weight-based DCS dosing will be measured by blood draws at several time points throughout iTBS treatment. Specifically, a pharmacokinetic curve will be generated on Day 1 of iTBS treatment from D-Cycloserine levels obtained at 6 timepoints; pre-ingestion, +30 mins, + 60 mins, + 90mins, +120mins and +24 hrs. Additional time points will be obtained prior to and 120 minutes after the fifth dose (Day 5 of TMS) and prior to and 120 minutes after the sixth dose (Day 6 of TMS, corresponding to the beginning of the second week of TMS).

Antidepressant effects will be quantified using the Montgomery Asberg Depression Rating Scale, a gold standard clinician rated instrument. Participants will complete a short battery of cognitive tests at the beginning and end of the study. Blood work and echocardiogram will be repeated after 4 weeks to confirm safety of low-dose DCS.

Participants will return to the lab for a follow-up assessment 4 weeks after they have finished the TMS protocol (week 8).

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 18 to 65 years
2. are competent to consent to treatment
3. have a confirmed diagnosis of DSM-5 criteria Major Depressive Disorder with a current episode of at least moderate severity of depression, single or recurrent
4. have failed to achieve a clinical response to one adequate trial of antidepressant medication within the current episode, or been unable to tolerate antidepressant medications.
5. have current episode of at least moderate severity of depression, as defined by a score ≥ 18 on the HAMD-17 item
6. have had no change in dose, or initiation of any psychotropic medication in the 4 weeks prior to randomization
7. are able to adhere to the treatment schedule
8. pass the TMS adult safety screening (TASS) questionnaire
9. have had blood work (complete blood count, electrolytes, BUN, creatinine, eGFR, AST, ALT and GGT, and ECG) within the reference range. Female participants must have a negative pregnancy test.

Exclusion Criteria:

1. Allergy to cycloserine.
2. have failed adequate trials of ≥4 antidepressant treatments in the current episode.
3. have an alcohol or substance use disorder within the last 3 months
4. have suicidal ideation (score of 4 ≥ on item 10 of MADRS)
5. are at a significant risk of harm to themselves or others
6. current symptoms of psychosis
7. history of psychosis
8. are currently pregnant, breast feeding or plan to become pregnant over the duration of the study
9. have a diagnosis of other primary psychiatric diagnoses as assessed by a study investigator to be primary and causing greater impairment than Major Depressive Disorder.
10. have failed a course of ECT in the current episode. Previous ECT treatment outside of the current episode does not influence inclusion.
11. history of non-response to TMS treatment.
12. have any significant neurological disorder or insult including, but not limited to: any condition likely to be associated with increased intracranial pressure, space occupying brain lesion, any history of epilepsy, cerebral aneurysm, Parkinson's disease, Huntington's chorea, multiple sclerosis, significant head trauma with loss of consciousness for greater than or equal to 5 minutes
13. have concomitant major unstable medical illness, cardiac pacemaker or implanted medication pump
14. have an intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed
15. if participating in psychotherapy, must have been in stable treatment for at least 3 months prior to entry into the study, with no anticipation of change in the frequency of therapeutic sessions, or the therapeutic focus over the duration of the study
16. are currently (or in the last 4 weeks) taking any benzodiazepine, cyclopyrrolone, gabapentin/pregabalin or anticonvulsant due to the potential to limit TMS efficacy
17. have an exclusion criteria for MRI: Those with a history of cranial, thoracic or abdominal surgery, with pacemakers, artificial joints or other metallic implants will be excluded from the MRI scan. Subjects that have agreed to participate in the MRI portion of the study will be pre-screened for any potential metal fragments in the body (particularly in the orbits) if they have had any history of doing metal work or have been involved in use/deployment of ammunitions/explosives, welding, piping etc).
18. are being currently treated with ethionamide or isoniazid (contraindicated with D-cycloserine)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) | Administered at baseline, at the halfway point (week 2), after rTMS treatment (week 4), and at one month follow up (week 8)
  Change in severity of depressive symptoms as measured by the MADRS, a clinician-rated instrument. The MADRS is a ten-item diagnostic questionnaire used to measure the severity of depressive episodes. The overall score ranges from 0 - 60. Cutoff points are 0-6 = normal, 7-9 = mild depression, 20-34 = moderate depression, >34 = severe depression.
Individual differences in D-cycloserine serum concentration will be correlated with clinical outcomes | 10 blood samples: PK curve over the first 2 days of TMS treatment (6 draws) and prior to ingestion and after 120 minutes on day 5 and day 6
  Examine whether differential change in clinical outcomes will be mediated by D-Cycloserine plasma levels following weight-based dosing. Participants will provide 10 blood samples to characterize plasma levels of D-Cycloserine following a weight-based dose. The primary efficacy measures will be examined in relation to drug blood levels.
Individual fidelity to the protocol will be correlated with differential change in primary outcomes | Daily Monday-Friday throughout study (4 weeks)
  All participants will be instructed to take the blinded capsule 90 - 120 minutes prior to TMS treatment, ensuring adequate time for drug absorption. Daily logs will be kept by the study staff to confirm time of capsule ingestion and TMS treatment. Any TMS sessions missed, capsule doses missed and/or capsule doses taken at the incorrect time will be tracked. The primary efficacy measures will be examined in relation to adherence to the protocol (20/20 TMS session completed with oral capsule taken between 90 - 120 minutes prior).
The variance in D-cycloserine level will be greater in the 100mg dosing condition than in the weight-based dosing condition. | PK curve done at baseline (fixed dose) and Day 1 of TMS (weight-based dose). Samples at pre-ingestion, +30 minutes, +60 minutes, +90 minutes, +120 minutes, and +24hours.
  The maximum serum concentration of D-cycloserine in blood serum will be measured by taking blood samples at various timepoints following oral D-cycloserine. Maximum serum concentration following 100mg oral D-cycloserine and weight-based oral D-cycloserine (dosed 25mg/17.5kg) will be compared. Blood samples will be drawn at baseline (pre-ingestion), +30 minutes, +60 minutes, +90 minutes and +24hours after a uniform dosing of 100mg of D-cycloserine and after a weight-based dosing of 25mg D-cycloserine per 17.5kg of body weight.
Determine whether blood serum levels of D-cycloserine achieved by weight-based dosing is consistent across time. | Day 1 of TMS, Day 5 of TMS, and Day 6 of TMS.
  Serum concentrations of weight-based oral D-cycloserine (dosed 25mg/17.5kg body weight) will be described by collecting blood samples 120 minutes after ingestion of the first, fifth and sixth dose.

SECONDARY OUTCOMES:
Number of participants that achieve clinical remission of depression | Administered at baseline, halfway (week 2), after rTMS treatment (week 4), and at one month follow up (week 8)
  Clinical remission of depressive symptoms will be measured by the Montgomery-Asberg Depression Rating Scale (MADRS); a clinician-rated instrument. The MADRS is a ten-item diagnostic questionnaire used to measure the severity of depressive episodes. The overall score ranges from 0 - 60. A score of </= 10 on the MADRS indicates clinical remission.
Number of participants that achieve clinical response (>=50% improvement in depression) | Administered at baseline, halfway (week 2), after rTMS treatment (week 4), and at one month follow up (week 8)
  Clinical depression response will be measured by the Montgomery-Asberg Depression Rating Scale (MADRS); a clinician-rated instrument. The MADRS is a ten-item diagnostic questionnaire used to measure the severity of depressive episodes. The overall score ranges from 0 - 60. A reduction of >/= 50% in the MADRS score indicates clinical response.
Changes in self-reported depression as measured by the Quick Inventory of Depressive Symptoms (QIDS-SR) | Administered at baseline, halfway (week 2), after rTMS treatment (week 4), and at one month follow up (week 8)
  The Quick Inventory of Depressive Symptomatology (QIDS) rates depression symptoms via self-assessment.Severity of depression can be judged based on the total score.
  1-5 = No depression 6-10 = Mild depression 11-15 = Moderate depression 16-20 = Severe depression 21-27 = Very severe depression
Changes in self-reported anxiety as measured by the Generalized Anxiety Disorder (GAD-7) questionnaire | Administered at baseline, halfway (week 2), after rTMS treatment (week 4), and at one month follow up (week 8)
  Anxiety symptoms will be assessed using the 7 item Generalized Anxiety Disorder (GAD-7) questionnaire. The GAD-7 measures self-reported feelings of anxiety within the last 2 weeks. Scores range from 0-21. Scores of 5, 10, and 15 represent cut points for mild, moderate, and severe anxiety, respectively.
Change in suicidal intentions | Administered at baseline, halfway (week 2), after rTMS treatment (week 4), and at one month follow up (week 8)
  The Scale for Suicide Ideation (SSI) is a brief 19-item scale that assesses the person's current intensity of attitudes, plans, and behaviors to commit suicide. Each question has 3 answer choices. The answer choice suggesting the least suicide intentions is scored as 0, and answer choice suggesting the most suicide intentions are scored as 2.
  Total score is determined based on the sum of all individual scores.
Change in Cognitive Function - THINC-integrated tool (THINC-it)- Choice Reaction Time | Administered at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  Cognitive function will be assessed using the THINC-it brief cognitive assessment tool. THINC-it includes a summation of four objective cognitive tests and a subjective cognitive questionnaire.
  The first objective cognitive test is called "spotter" and measures choice reaction time by calculating the total time that elapses between the presentation of a stimulus and the occurrence of a response in a task that requires a participant to make one of two different responses depending on which stimuli is presented. Less time between presentation of stimulus and occurrence of a response can be used as an indicator for better reaction time.
  Total results from the THINC-it assessment indicate cognitive performance compared to healthy age-, sex- and education-matched individuals. Change between the two arms will be assessed.
Change in Cognitive Function - THINC-integrated tool (THINC-it)- Working Memory | Administered at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  Cognitive function will be assessed using the THINC-it brief cognitive assessment tool. THINC-it includes a summation of four objective cognitive tests and a subjective cognitive questionnaire.
  The second objective cognitive test is called "Symbol Check" and is an n-back test. N-back tests measure working memory by presenting the subject with a sequence of stimuli, and the task consists of selecting the stimuli that was presented n steps earlier in the sequence. The greater amount of correct responses can be used as an indicator of better working memory.
  Total results from the THINC-it assessment indicate cognitive performance compared to healthy age-, sex- and education-matched individuals. Change between the two arms will be assessed.
Change in Cognitive Function - THINC-integrated tool (THINC-it)- Digit Symbol Substitution | Administered at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  Cognitive function will be assessed using the THINC-it brief cognitive assessment tool. THINC-it includes a summation of four objective cognitive tests and a subjective cognitive questionnaire.
  The third objective cognitive test is called "CodeBreaker" and is a Digit Symbol Substitution Test (DSST). DSST involves a key consisting of the numbers 1-6, each paired with a unique symbol. Below the key are a series of the numbers 1-6 in random order and repeated several times. Subjects must select the corresponding symbol as fast as possible. The number of correct symbols within the allowed time is measured, with higher number of correct symbols indicating greater cognitive function.
  Total results from the THINC-it assessment indicate cognitive performance compared to healthy age-, sex- and education-matched individuals. Change between the two arms will be assessed.
Change in Cognitive Function - THINC-integrated tool (THINC-it)- Trail Making Test part B | Administered at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  Cognitive function will be assessed using the THINC-it brief cognitive assessment tool. THINC-it includes a summation of four objective cognitive tests and a subjective cognitive questionnaire.
  The fourth objective cognitive test is called "Trails" and is a version of the Trail Making Test part B (TMT-B). The subject is presented with numbers and letters in circles placed in random array on the screen. The subject must draw a line from one circle to the next in ascending order; however, s/he must alternate the circles with numbers in them and circles with letters in them (ie, 1-A-2-B-3-C etc). The TMT is a timed test and the goal is to complete the tests accurately and as quickly as possible. Less time to accurately complete the trial indicates greater cognitive function.
  Total results from the THINC-it assessment indicate cognitive performance compared to healthy age-, sex- and education-matched individuals. Change between the two arms will be assessed.
Implicit Suicidality | Administered at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  Death Implicit Association Test (D-IAT) is a behavioral test that measures the strength of automatic (implicit) associations between concepts in people's minds relying on latency measures in a simple sorting task. The strength of an association between concepts of "death" and "ones self" is measured by the standardized mean difference score of the 'hypothesis-inconsistent' pairings and 'hypothesis-consistent' pairings
Clinical Global Impression- Severity | Administered at baseline, halfway (week 2), after rTMS treatment (week 4), and at one month follow up (week 8)
  The CGI-Severity scale is clinician rated from 1-7 representing 'Not at all ill' to 'Severely ill'.
Clinical Global Impression- Improvement | Administered at baseline, halfway (week 2), after rTMS treatment (week 4), and at one month follow up (week 8)
  The CGI-Improvement scale is a clinician rated 1-7, representing the range between 'Very much improved' and 'Very much worse' from the baseline visit.
Improvements in depressive symptoms will persist until the 8 week timepoint | Administered at baseline, halfway (week 2), after rTMS treatment (week 4), and at one month follow up (week 8)
  Change in severity of depressive symptoms as measured by the MADRS, a clinician-rated instrument. The MADRS is a ten-item diagnostic questionnaire used to measure the severity of depressive episodes. The overall score ranges from 0 - 60. Cutoff points are 0-6 = normal, 7-9 = mild depression, 20-34 = moderate depression, >34 = severe depression.
Change in Cognitive Function - THINC-integrated tool (THINC-it)- Perceived Deficits Questionnaire - 5 item scale (PDQ-5) | Administered at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  Cognitive function will be assessed using the THINC-integrated tool (THINC-it) brief cognitive assessment tool. THINC-it includes a summation of four objective cognitive tests and a subjective cognitive questionnaire.
  The cognitive questionnaire is called the Perceived Deficits Questionnaire - 5 item scale (PDQ-5). The questionnaire assesses self perceived cognition by asking questions about attention/concentration, retrospective memory, prospective memory, and planning/organization. Each item is rated on a 5-point scale ranging from 0 (never) to 5 (almost always). Higher scores indicate greater perceived deficits in cognition.
  Total results from the THINC-it assessment indicate cognitive performance compared to healthy age-, sex- and education-matched individuals. Change between the two arms will be assessed.

OTHER OUTCOMES:
Side Effects | Administered at baseline, after rTMS treatment (week 4), and at one month follow up (week 8)
  Side effects will be tracked through the Toronto Side Effects Scale (TSES). The TSES is a self reported questionnaire that assesses incidence, frequency, and severity of central nervous system, gastrointestinal, and sexual side effects. Individuals will be asked to rate frequency of each symptom within the last week on a 5-point scale, from "Never" (1) to "Everyday" (5). Severity of each symptom is similarly rated on a 5-point scale, from "No trouble" (1) to "Extreme Trouble" (5). Total score from the Toronto Side Effect Scale will be analyzed using paired t-test.
Incidence of Treatment-Emergent Adverse Events | Daily Monday-Friday throughout study (4 weeks) and at one month follow up
  Adverse events will be tracked and recorded. Adverse events will not occur at a higher rate than is expected for iTBS.
Safety hypothesis: There will be no clinically significant changes in bloodwork; Sodium level | Baseline and after rTMS treatment (week 4)
  An electrolyte panel will be used to measure the amount of sodium present in the blood from a whole blood sample, measured in mmol/L. Results must be within normal reference range prior to entering the study. Results from baseline and treatment end will be compared with paired t-tests.
Safety hypothesis: There will be no clinically significant changes in bloodwork; Potassium level | Baseline and after rTMS treatment (week 4)
  An electrolyte panel will be used to measure the amount of potassium present in the blood from a whole blood sample, measured in mmol/L. Results must be within normal reference range prior to entering the study. Results from baseline and treatment end will be compared with paired t-tests.
Safety hypothesis: There will be no clinically significant changes in bloodwork; Chloride level | Baseline and after rTMS treatment (week 4)
  An electrolyte panel will be used to measure the amount of chloride present in the blood from a whole blood sample, measured in mmol/L. Results must be within normal reference range prior to entering the study. Results from baseline and treatment end will be compared with paired t-tests.
Safety hypothesis: There will be no clinically significant changes in bloodwork; Hemoglobin | Baseline and after rTMS treatment (week 4)
  A complete blood count (CBC) panel will be used to measure the amount of hemoglobin present in the blood from a whole blood sample, measured in g/L. Results must be within normal reference range prior to entering the study. Results from baseline and treatment end will be compared with paired t-tests.
Safety hypothesis: There will be no clinically significant changes in bloodwork; Hematocrit | Baseline and after rTMS treatment (week 4)
  A complete blood count (CBC) panel will be used to measure the amount of hematocrit present in the blood from a whole blood sample, measured in L/L. Results must be within normal reference range prior to entering the study. Results from baseline and treatment end will be compared with paired t-tests.
Safety hypothesis: There will be no clinically significant changes in bloodwork; White Blood Cell count | Baseline and after rTMS treatment (week 4)
  A complete blood count (CBC) panel will be used to measure the amount of white blood cells (WBC) present in the blood from a whole blood sample, measured in 10^9/L. Results must be within normal reference range prior to entering the study. Results from baseline and treatment end will be compared with paired t-tests.
Safety hypothesis: There will be no clinically significant changes in bloodwork; Red Blood Cell count | Baseline and after rTMS treatment (week 4)
  A complete blood count (CBC) panel will be used to measure the amount of red blood cells (RBC) present in the blood from a whole blood sample, measured in 10^12/L. Results must be within normal reference range prior to entering the study. Results from baseline and treatment end will be compared with paired t-tests.
Safety hypothesis: There will be no clinically significant changes in bloodwork; platelets | Baseline and after rTMS treatment (week 4)
  A complete blood count (CBC) panel will be used to measure the amount of platelets present in the blood from a whole blood sample, measured in 10^9/L. Results must be within normal reference range prior to entering the study. Results from baseline and treatment end will be compared with paired t-tests.
Safety hypothesis: There will be no clinically significant changes in bloodwork; AST | Baseline and after rTMS treatment (week 4)
  An AST test measures the level of aspartate aminotransferase (AST) present in the blood from a whole blood sample, measured in U/L. Results must be within normal reference range prior to entering the study. Results from baseline and treatment end will be compared with paired t-tests.
Safety hypothesis: There will be no clinically significant changes in bloodwork; ALT | Baseline and after rTMS treatment (week 4)
  An ALT test measures the level of alanine transaminase (ALT) present in the blood from a whole blood sample, measured in U/L. Results must be within normal reference range prior to entering the study. Results from baseline and treatment end will be compared with paired t-tests.
Safety hypothesis: There will be no clinically significant changes in bloodwork; GGT | Baseline and after rTMS treatment (week 4)
  A GGT test measures the level of gamma-glutamyl transpeptidase (GGT) present in the blood from a whole blood sample, measured in U/L. Results must be within normal reference range prior to entering the study. Results from baseline and treatment end will be compared with paired t-tests.
Safety hypothesis: There will be no clinically significant changes in bloodwork; BUN | Baseline and after rTMS treatment (week 4)
  A BUN test (aka blood urea nitrogen test) measures the level of urea nitrogen present in the blood from a whole blood sample, measured in mmol/L. Results must be within normal reference range prior to entering the study. Results from baseline and treatment end will be compared with paired t-tests.
Safety hypothesis: There will be no clinically significant changes in bloodwork; Creatinine | Baseline and after rTMS treatment (week 4)
  A creatinine blood test measures the level creatinine present in the blood from a whole blood sample, measured in umol/L. Results must be within normal reference range prior to entering the study. Results from baseline and treatment end will be compared with paired t-tests.
Safety hypothesis: There will be no clinically significant changes in bloodwork; eGFR | Baseline and after rTMS treatment (week 4)
  In adults, glomerular filtration rate can be easily estimated using the CKD-EPI GFR equation.
  This formula uses the patient's age and gender with the measured blood creatinine value to estimate glomerular filtration rate, or eGFR. eGFR is measured in mL/min/1.73m^2.
  Results must be within normal reference range prior to entering the study. Results from baseline and treatment end will be compared with paired t-tests.
Safety hypothesis: There will be no clinically significant changes in QTc | Baseline and after rTMS treatment (week 4)
  Electrical activity of the heart will be measured by an electrocardiogram (ECG). The QT interval is calculated as the time from the start of the Q wave to the end of the T wave. The QT interval is corrected for heartrate (QTc), a process performed automatically by modern ECG recorders. Results must be within normal range prior to entering the study. QTc from baseline to treatment end will be compared with paired t-tests.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander McGirr, MD PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No